CLINICAL TRIAL: NCT05155098
Title: 2 Years Prospective Study to Collect Real-life Data On the Retention, Quality of Life, Effectiveness and Treatment Pattern of Secukinumab in Adult Patients With Moderate to Severe Plaque Psoriasis, Psoriatic Arthritis, Ankylosing Spondylitis and Non-radiographic Axial spondyloarthriTis (PROMPT)
Brief Title: 2 Years Prospective Study to Collect Real-life Data on the Retention, Quality of Life, Effectiveness and Treatment Pattern of Secukinumab in Adult Patients With Moderate to Severe Plaque Psoriasis, Psoriatic Arthritis, Ankylosing Spondylitis and Non-radiographic Axial Spondyloarthritis
Acronym: PROMPT
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457ATH02
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Moderate to Severe Plaque Psoriasis; Psoriatic Arthritis; Ankylosing Spondylitis; Non-radiographic Axial Spondyloarthritis
Keywords: Moderate to severe plaque psoriasis; Psoriatic arthritis; Ankylosing spondylitis; Non-radiographic axial spondyloarthritis; NIS; Thailand; secukinumab
MeSH Terms: conditions — Arthritis, Psoriatic; Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- secukinumab: Patients receiving secukinumab in real world practice
  Interventions: Other: secukinumab

INTERVENTIONS:
Other: secukinumab — Prospective observational study. There is no treatment allocation. Patients who are receiving or intend to receive secukinumab are eligible to enroll into this study.

SUMMARY:
This is an observational, prospective primary data collection study. The duration of observation is 2 years after study enrolment date. Disease and treatment history will be retrospectively reviewed from medical record at enrollment with no time limits for the key diagnosis of enrolment (plaque psoriasis, psoriatic arthritis, ankylosing spondylitis and non-radiographic axial spondyloarthropathy).

DETAILED DESCRIPTION:
After the baseline visit, data will be collected for each patient prospectively every 6 months for up to 2 years. At each visit, effectiveness parameters, as well as the patients' QoL and treatment pattern will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent of the patient to participate in the study
2. Age 18-80 years.
3. Patients with an assured diagnosis by the treating physician of active moderate to severe plaque psoriasis or active PsA or active AS or active non-radiographic axial SpA.
4. Patients must have received the official approval to receive secukinumab in Dermatology Disease Prior Authorization (DDPA) or Rheumatology Disease Prior Authorization (RDPA) before study participation or the decision to treat patient's condition with secukinumab is happened before entering the study
5. Patients must receive the first dose of secukinumab during the study enrollment period.
6. Patients for whom the decision for a therapy with secukinumab is made by the attending treating physician, regardless of this non-interventional study.
7. Patients who have EQ-5D score before start the 1st dose secukinumab.

Exclusion Criteria:

1. Any medical or psychological condition in the treating physician's opinion which may prevent the patient from study participation for the 2 year study period.*
2. Patients participating in parallel in other interventional clinical trial.
3. Patients participated in an interventional clinical trial with secukinumab involvement in the past.

   * Note: For example, patients diagnosed with a terminal illness and those with cognitive impairment due to dementia and Alzheimer's disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderate to severe plaque psoriasis, psoriatic arthritis, ankylosing spondylitis and non-radiographic axial spondyloarthritis
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Retention rate of secukinumab therapy | 2 years
  Retention rate is defined as percentage of patients who have not discontinued the medication.

SECONDARY OUTCOMES:
Retention rate of secukinumab therapy by individual indication | year 1, year 2
  Retention rate is defined as percentage of patients who have not discontinued the medication.
Change in QoL by EQ-5D Visual Analog Scale (VAS) | Baseline, month 6, month 12, month 18, month 24
  Euro-QoL-5 Dimension Questionnaire (EQ-5D) is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.
Treatment pattern | Month 6, month 12, month 18, month 24
  Proportion of patients for each indication with alterations of secukinumab treatment regimen and reasons for.
Work/school absenteeism | 2 years
  Number of days of absenteeism from work/school due to health condition during each visit. Health condition which is considered to be related to the absenteeism will be determined by the treating physicians on the relationship with psoriasis, psoriatic arthritis or non-radiographic axial SpA or others conditions.
Patients with Psoriasis: Proportions of patients achieving a PASI 75, 90, and 100 responses | Month 6, month 12, month 18, month 24
  Psoriasis Area and Severity Index (PASI) takes into account the extent of the disease, as well as the severity of erythema, scaling, and thickness in different body areas affected by psoriasis.
  * A PASI 75 represents an improvement in the PASI score of at least 75% as compared with baseline.
  * A PASI 90 represents an improvement in the PASI score of at least 90% as compared with baseline.
  * A PASI 100 response corresponds to complete clearing of psoriasis (PASI = 0).
Patients with Psoriasis: Changes between PASI response categories over time | 2 Years
  Changes between PASI response categories over time after starting participation in the study to be collected.
Patients with Psoriasis: Absolute PASI scores | Month 6, month 12, month 18, month 24
  Absolute PASI scores to be collected
Patients with Psoriasis: Changes in absolute and relative PASI scores over time | Baseline, month 6, month 12, month 18, month 24
  Relative PASI, also called PASI response, is reported as a percent change from baseline PASI.
  Absolute PASI is reported as a score to reflect the current status of severity of disease.
Patients with Psoriasis: Proportion of patients achieving a PGA 0/1 response | Month 6, month 12, month 18, month 24
  Physician Global Assessment (PGA) 0/1 response = clear/almost clear skin
Patients with Psoriasis: Proportion of patients achieving a DLQI 0/1 response | Month 6, month 12, month 18, month 24
  Dermatology Life Quality Index (DLQI) is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such psoriasis. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) 1 ( a little) to 3 (very much). "Not relevant" is a valid score also and is scored as 0.
Patients with Psoriasis: Correlation between PASI and DLQI score | 2 years
  Correlation analysis will be performed using Pearson's correlation or Spearman's correlation, depending on normality.
Patients with Psoriatic Arthritis: 78 TJC and 76 SJC | 1 year, 2 years
  78 tender joint count (TJC) is determined by physical examination of 78 joint counts that are assessed for tenderness.
  76 swollen joint count (SJC) is determined by physical examination of 76 joint counts that are classified as either swollen or not swollen.
Patients with Psoriatic Arthritis: Physician's global assessment (PGA) | 1 year, 2 years
  VAS scale will be used to measure disease activity. The Visual Analog Scale (VAS) is a commonly used measurement of pain, discomfort, that goes from 0 meaning no pain to 100 meaning worst imaginable pain
Patients with Psoriatic Arthritis: Total patient pain assessed by visual analog scale (VAS) | 1 year, 2 years
  The Visual Analog Scale (VAS) is a commonly used measurement of pain, discomfort, that goes from 0 meaning no pain to 100 meaning worst imaginable pain
Patients with Psoriatic Arthritis: Presence of any dactylitis | 1 year, 2 years
  Dactylitis is severe inflammation of the finger and toe joints.
Patients with Psoriatic Arthritis: Presence of any enthesitis | 1 year, 2 years
  Presence of any enthesitis in the following sites: lateral epicondyle humerus left and right, Achilles left and right and medial condyle femur left and right.
  Enthesitis refers to inflammation of entheses, the site where ligaments or tendons insert into the bones.
Patients with Psoriatic Arthritis: Appearance of new bone erosions or worsening of pre-existing erosions | 1 year, 2 years
  Appearance of new bone erosions or worsening of pre-existing erosions in the hands and feet by X-ray assessment, according to the Treating Physician's opinion
Patients with Psoriatic Arthritis: Proportion of patients achieving a PASI 75, 90, and 100 response | month 6, month 12, month 18 and month 24
  Psoriasis Area and Severity Index (PASI) takes into account the extent of the disease, as well as the severity of erythema, scaling, and thickness in different body areas affected by psoriasis.
  * A PASI 75 represents an improvement in the PASI score of at least 75% as compared with baseline.
  * A PASI 90 represents an improvement in the PASI score of at least 90% as compared with baseline.
  * A PASI 100 response corresponds to complete clearing of psoriasis (PASI = 0).
Patients with Psoriatic Arthritis: Changes between PASI response categories over time | 2 years
  Changes between PASI response categories over time after starting participation in the study
Patients with Psoriatic Arthritis: Absolute PASI scores | month 6, month 12, month 18 and month 24
  Absolute PASI scores to be collected
Patients with Psoriatic Arthritis: Changes in absolute and relative PASI scores over time | 2 years
  Changes in absolute and relative PASI scores over time after inclusion into the study.
Patients with Psoriatic Arthritis: Changes of HAQ-DI score | month 6, month 12, month 18 and month 24
  Health Assessment Questionnaire Disability Index (HAQ-DI) assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in 8 categories of functioning including dressing, rising, eating, walking, hygiene, reach, grip and usual activities. The stem of each item asks 'Over the past week, "are you able to..." perform a particular task'. Each item is scored on a 4 point scale from 0 - 3, representing normal, no difficulty (0), some difficulty (1), much difficulty (2) and unable to do (3). The disability index score is calculated as the mean of the available category scores, ranging from 0 to 3. A negative change from baseline indicates improvement.(Only at sites where HAQ-DI score is part of clinical routine).
Patients with Psoriatic Arthritis: Changes of FACIT-Fatigue score | month 6, month 12, month 18 and month 24
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) assesses self-reported fatigue and its impact upon daily activities and function.
  FACIT-Fatigue Scale: overall score (0 to 52)=the sum of scores for 13 questions. For each question, par. rated their condition for the past week on a 5-point scale: 0 (not at all) to 4 (very much). A high score indicates low fatigue.
  (Only at sites where FACIT-Fatigue score is part of clinical routine).
Patients with Psoriatic Arthritis: Correlation between effectiveness measures, HAQ-DI, and FACIT-Fatigue scores | 2 years
  Correlation analysis will be performed using Pearson's correlation or Spearman's correlation, depending on normality.
Patients with Ankylosing spondylitis: Bath AS disease activity index (BASDAI) response | year 1, year 2
  BASDAI is a participant-reported assessment consisting of 6 questions that relate to 5 major symptoms relevant to ankylosing spondylitis: 1) Fatigue, 2) Spinal pain, 3) Peripheral arthritis, 4) Enthesitis, 5) Intensity, and 6) Duration of morning stiffness. Participants need to score each item with a score from 0 to 10. Total score is obtained from the average of symptom scores ranging 0 (no problem) to 10 (worst problem), with a higher score indicating more severe symptoms.
Patients with Ankylosing spondylitis: Patient's global assessment of disease activity | year 1, year 2
  Patient's global assessment of disease activity will be measured using VAS scale or NRS (numeric rating scale). NRS scale goes from 0 to 10 (0= no activity, 10= activity)
Patients with Ankylosing spondylitis: C-reactive protein (CRP) or high-sensitivity CRP (hsCRP) | year 1, year 2
  CRP or high-sensitivity CRP to be collected
Patients with Ankylosing spondylitis: Total spinal pain assessed using VAS scale | year 1, year 2
  The Visual Analog Scale (VAS) is a commonly used measurement of pain, discomfort, that goes from 0 meaning no pain to 100 meaning worst imaginable pain
Patients with Ankylosing spondylitis: Presence of any enthesitis | 2 years
  Presence of any enthesitis in the following sites:
  * Costochondral 1 right/left
  * Costochondral 7 right/left
  * Spina iliaca anterior superior right/left
  * Crista iliaca right/left
  * Spina iliaca posterior right/left
  * Processus spinosus L5
  * Achilles tendon, insertion right/left Enthesitis refers to inflammation of entheses, the site where ligaments or tendons insert into the bones.
Patients with Ankylosing spondylitis: Appearance or worsening of lesions at anterior sites of the vertebrae assessed by X-ray | year 1, year 2
  Appearance or worsening, according to the treating physician's opinion, of any of the following lesions at anterior sites of the vertebrae assessed by X-ray (when available):
  * Squaring
  * Erosions
  * Sclerosis
  * Syndesmophytes
  * Bridging syndesmophytes
Patients with Ankylosing spondylitis: Appearance or worsening of bone marrow edema (BME) in the spine and/or sacro-iliac joints assessed by magnetic resonance imaging (MRI) | year 1, year 2
  Appearance or worsening (according to the Treating Physician's opinion) of bone marrow edema (BME) in the spine and/or sacro-iliac joints assessed by magnetic resonance imaging (MRI) (when available).
Ankylosing spondylitis and non-radiographic axial SpA: Changes of FACIT-Fatigue score compared to baseline | month 6, month 12, month 18 and month 24
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) assesses self-reported fatigue and its impact upon daily activities and function.
  FACIT-Fatigue Scale: overall score (0 to 52)=the sum of scores for 13 questions. For each question, par. rated their condition for the past week on a 5-point scale: 0 (not at all) to 4 (very much). A high score indicates low fatigue.
Ankylosing spondylitis: Correlation between ASDAS, BASDAI, and FACIT-Fatigue scores | 2 years
  Data from BASDAI, patient's global assessment (NRS) and CRP/hsCRP can be used to calculate the AS disease activity score (ASDAS).
  Correlation analysis will be performed using Pearson's correlation or Spearman's correlation, depending on normality.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Thailand (7):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Muang, Thailand
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Kaen
  - Novartis Investigative Site, Nakhon Ratchasima

IPD SHARING:
Plan to Share IPD: No